CLINICAL TRIAL: NCT04055038
Title: Randomized Phase II/III Trial to Assess the Efficacy of Platinum-based Chemotherapy vs Standard Non-platinum Therapy in Patients With Platinum-resistant Recurrent Ovarian Cancer (ROC)
Brief Title: Efficacy of Platinum-based Chemotherapy in Platinum-resistant Ovarian Cancer) (EPITOC)
Acronym: EPITOC
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Blokhin's Russian Cancer Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROC2019
Record Dates: First submitted 2019-04-28; First posted 2019-08-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Ovarian Cancer; Ovarian Neoplasms; Serous Adenocarcinoma; BRCA1 Mutation; BRCA2 Mutation; Chemotherapy
MeSH Terms: conditions — Ovarian Neoplasms; Cystadenocarcinoma, Serous

STUDY DESIGN:
Intervention Model Description: Randomized phase II/III trial to assess the efficacy of platinum-based chemotherapy vs standard non-platinum therapy in patients with platinum-resistant recurrent ovarian cancer (ROC)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platinum-based chemotherapy (Experimental): This is an experimental arm of this study. Allowed therapeutic options:
  1. Paclitaxel 60-80 mg/m2 + carboplatin area under curve (AUC) 2-2.7 d 1, 8, 15 every 3 or 4 weeks (Q3W or Q4W);
  2. Gemcitabine 1000 mg/m2 d 1, 8 + cisplatin 75 mg/m2 1 every 3 weeks;
  3. Doxorubicin 40-50 mg/m2 d 1 + carboplatin AUC5 or cisplatin 60-75 mg/m2 d 1 every 3 weeks;
  4. Topotecan 0.75 mg/m2 d 1-3 + cisplatin 60-75 mg/m2 or carboplatin AUC 4-5 d 1 every 3 weeks;
  5. Etoposide 100 mg once daily orally d 1-7 + cisplatin 60-75 mg/m2 d1 every 3 weeks.
  Up to 6 cycles of chemotherapy will be administered to study participants allocated to this arm.
  Interventions: Drug: Platinum-Based Drug
- Non-platinum monochemotherapy (Active Comparator): This is a control arm of this study. Allowed therapeutic options:
  1. Paclitaxel 60-80 mg/m2 weekly (or day 1, 8, 15 every 4 weeks schedule);
  2. Gemcitabine 1000 mg/m2 d 1, 8, 15 every 4 weeks;
  3. Doxorubicin 50-60 mg/m2 d 1 every 3 weeks;
  4. Topotecan 1,2-1,5 mg/m2 d 1-5 every 3 weeks;
  5. Etoposide 100 mg once daily orally d 1-10 every 3 weeks.
  Up to 6 cycles of chemotherapy will be administered to study participants allocated to this arm.
  Interventions: Drug: Conventional chemotherapy

INTERVENTIONS:
Drug: Platinum-Based Drug — Reintroduction of platinum-based chemotherapy
  Arms: Platinum-based chemotherapy
Drug: Conventional chemotherapy — Conventional chemotherapy
  Arms: Non-platinum monochemotherapy

SUMMARY:
This is a phase II/III randomized controlled trial to evaluate efficacy of platinum-based chemotherapy vs conventionally prescribed non-platinum monochemotherapy in patients with platinum-resistant ovarian cancer

DETAILED DESCRIPTION:
Recurrent ovarian cancer (ROC) is usually subdivided to platinum-sensitive (platinum-free interval [PFI] ≥6 mo.) and platinum-resistant ovarian cancer [PROC] (PFI <6 mo.) subtypes. Prognosis for the latter group is dismal and current guidelines recommend treating these patients with non-platinum based chemotherapy. However, the evidence behind this is quite unconvincing and according to recent data patients with non-platinum refractory platinum-resistant ovarian cancer could derive benefit from platinum rechallenge. This trial is designed for head-to-head comparison of platinum and non-platinum therapy efficacy in treatment of platinum-resistant ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years;
* Histologically confirmed epithelial ovarian cancer (excluding mucinous, clear-cell and low-grade subtypes);
* Ovarian cancer recurrence within 3-6 months after completion of platinum-based chemotherapy (given to possible variability in follow-up practices and tumor growth kinetics patients with platinum-free interval ≥3 and <7 months will be considered platinum-resistant);
* Platinum-free interval ≤12 months;
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2;
* Response to penultimate platinum-based chemotherapy defined as partial or complete response assessed by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria or ≥50% reduction in CA-125 concentration for patients without measurable lesions;
* Not refractory to penultimate platinum-based chemotherapy regimen (ie, the disease did not progress during platinum-based chemotherapy and within ≤3 months after its completion);
* Patients received ≤3 lines of prior chemotherapy;
* No central nervous system (CNS) metastatic involvement;
* No severe and uncontrolled concomitant diseases;
* Adequate organ function:

  * Bone marrow - hemoglobin ≥ 90 g/l; Neutrophils ≥1,5x109/l; Platelets ≥75x109/l);
  * Renal - estimated creatinine clearance ≥50 ml/min (determined by Cockcroft-Gault equation);
  * Hepatic - alanine aminotransferase (ALaT) & aspartate transaminase (ASaT) ≤3 upper limit of normal (ULN), total bilirubin ≤ 25 umol/l;
* Known BRCA1/2 mutation status as it will be used for stratification;
* Life expectancy >3 months;
* Patient is willingly consent to participate in the trial and signed informed consent form

Exclusion Criteria:

* Platinum-refractory ovarian cancer defined as disease progression during penultimate platinum-based chemotherapy or ≤3 month after its completion;
* No response to penultimate platinum-based chemotherapy;
* Mucinous, clear-cell or low-grade serous/endometrioid histology;
* >3 lines of prior therapy lines for advanced ovarian cancer (prior maintenance endocrine therapy or poly ADP ribose polymerase (PARP) inhibitors is allowed);
* Prior therapy with PARP-inhibitors and endocrine therapy as a treatment for progressive ovarian cancer;
* Platinum-free interval >12 months;
* Symptoms of bowel obstruction of any etiology;
* Contraindications to platinum-based chemotherapy;
* Planned administration of PARP inhibitors during or after this line of chemotherapy;
* Life expectancy <3 months;
* Uncontrolled and/or severe concomitant diseases (eg, uncontrolled diabetes mellitus, renal failure, hepatic failure, uncontrolled arterial hypertension, arrhythmia, heart failure);
* Metastatic CNS involvement;
* Neuropathy grade >2.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — due to the nature of this disease only female participants are allowed
Enrollment: 164 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (RR) according to RECIST 1.1 criteria | 0-18 weeks
  Primary outcome for Phase II part: response rate to treatment according to RECIST1.1 criteria. For patients without measurable disease Rustin criteria is allowed.
Overall survival defined as time from randomization to death from any reason; | 1 year
  Primary outcome for Phase III part: 2. Overall survival defined as time from randomization to death from any reason

SECONDARY OUTCOMES:
Progression-free survival | 12 months
  Progression-free survival (PFS) defined as time from randomization to disease progression according to RECIST 1.1 criteria or death from any reason;
Overall survival | 12 months
  Overall survival defined as time from randomization to death from any reason (for Phase II part only);
Progression-free survival 2 (PFS2) | 24 months
  PFS2 defined as time from randomization to second disease progression event according to RECIST 1.1 criteria or death from any reason;
Objective response rate (RR) according to RECIST 1.1 criteria | 12 months
  Response rate to treatment according to RECIST1.1 criteria. For patients without measurable disease Rustin criteria is allowed (only for Phase II part).

CONTACTS AND LOCATIONS:
Locations (1):
- N.N. Blokhin Cancer Research Center, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No